CLINICAL TRIAL: NCT02505399
Title: TIcagrelor in Rotational Atherectomy to Reduce TROPonin Enhancement: the TIRATROP Study, a Randomized Controlled Trial
Brief Title: TIcagrelor in Rotational Atherectomy to Reduce TROPonin Enhancement
Acronym: TIRATROP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RC31/14/7445
Record Dates: First submitted 2015-06-03; First posted 2015-07-22 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2018-12

CONDITIONS: Atherosclerosis
Keywords: Rotational Atherectomy; clopidogrel; thrombosis; ticagrelor
MeSH Terms: conditions — Atherosclerosis; Thrombosis | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ticagrelor (Experimental): In the intervention group, Ticagrelor will be administered orally, according to the following scheme:
  * 180 mg the evening preceding (and at least 6 hours before) rotational atherectomy (Day -1),
  * 90 mg the following morning (D Day before rotational atherectomy and angioplasty),
  * 90 mg the following evening (D Day after rotational atherectomy and angioplasty),
  * 90 mg twice daily the day after the procedure of rotational atherectomy and angioplasty (Day +1).
  Interventions: Drug: ticagrelor
- clopidogrel (Active Comparator): In the control group, Clopidogrel will be administered orally, according to the following scheme:
  * 300 mg the evening preceding (and at least 6 hours before) rotational atherectomy (Day -1),
  * 75 mg the following morning (D Day before rotational atherectomy and angioplasty),
  * 0 mg the following evening (D Day after rotational atherectomy and angioplasty),
  * 75 mg once daily the day after the procedure of rotational atherectomy and angioplasty (Day +1).
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: ticagrelor — Ticagrelor will be administered orally, according to the following scheme:
  * 180 mg the evening preceding (and at least 6 hours before) rotational atherectomy (Day -1),
  * 90 mg the following morning (D Day before rotational atherectomy and angioplasty),
  * 90 mg the following evening (D Day after rotational atherectomy and angioplasty),
  * 90 mg twice daily the day after the procedure of rotational atherectomy and angioplasty (Day +1).
  Other Names: ticagrelor per os
  Arms: ticagrelor
Drug: clopidogrel — Clopidogrel will be administered orally, according to the following scheme:
  * 300 mg the evening preceding (and at least 6 hours before) rotational atherectomy (Day -1),
  * 75 mg the following morning (D Day before rotational atherectomy and angioplasty),
  * 0 mg the following evening (D Day after rotational atherectomy and angioplasty),
  * 75 mg once daily the day after the procedure of rotational atherectomy and angioplasty (Day +1).
  Other Names: clopidrogel per os
  Arms: clopidogrel

SUMMARY:
Rotational atherectomy (RA) prior to angioplasty is the reference treatment for highly calcified atherosclerotic coronary lesions. It aims at fragmenting calcium deposits into microscopic particulates to allow less hazardous coronary revascularization and stenting. The main drawback associated with the procedure is the subsequent enhancement of platelet aggregation which promotes the distal embolization of micro-thrombi and atherosclerotic fragments. In order to limit these complications, a double antiplatelet therapy is required (generally Clopidogrel + Aspirin) when RA procedures are performed. Clopidogrel inhibits the protein P2Y12 which is a cornerstone in platelet aggregation. Ticagrelor is a new antiplatelet agent that provides faster and greater P2Y12 inhibition than Clopidogrel. It is currently indicated to reduce risk of cardiovascular events in patients hospitalized for coronary revascularization after an acute coronary syndrome. Ticagrelor has never been evaluated so far in stable coronary patients treated with rotational atherectomy prior to angioplasty.

DETAILED DESCRIPTION:
Rotational atherectomy (RA) prior to angioplasty is the reference treatment for highly calcified atherosclerotic coronary lesions. It aims at fragmenting calcium deposits into microscopic particulates to allow less hazardous coronary revascularization and stenting. The main drawback associated with the procedure is the subsequent enhancement of platelet aggregation which promotes the distal embolization of micro-thrombi and atherosclerotic fragments. In order to limit these complications, a double antiplatelet therapy is required (generally Clopidogrel + Aspirin) when RA procedures are performed. Clopidogrel inhibits the protein P2Y12 which is a cornerstone in platelet aggregation. It is characterized by a slow and variable transformation of a prodrug into an active metabolite and by a remaining risk of thrombosis and myocardial infarction. Ticagrelor is a new antiplatelet agent that provides faster and greater P2Y12 inhibition than Clopidogrel. It is currently indicated to reduce risk of cardiovascular events in patients hospitalized for coronary revascularization after an acute coronary syndrome. Ticagrelor has never been evaluated so far in stable coronary patients treated with rotational atherectomy prior to angioplasty.

ELIGIBILITY:
Inclusion criteria :

* Stable coronary patient, or patient presenting with a non ST-elevation acute coronary syndrome without troponin elevation, or with troponin back to normal,
* Patient treated with a combination of Aspirin + Clopidogrel before hospitalization at the study center,
* Patient with at least one highly calcified coronary lesion eligible for rotational atherectomy prior to angioplasty,
* Patient agreed to participate after full information on the study.

Exclusion criteria :

* Acute coronary syndrome with ST-elevation,
* Plasma troponin level higher than 3 times the upper limit of the laboratory,
* Lesion located on a coronary bypass,
* Coronary thrombus diagnosed by angiography,
* Coronary dissection diagnosed by angiography,
* Left ventricular ejection fraction lower than 30%,
* Contra-indication to use Ticagrelor or Clopidogrel as listed in the Summary of Product Characteristics (SmPC, annex 1 & 2):

  * Known hypersensitivity to the active substance or to the excipients,
  * Active pathological bleeding,
  * History of intracranial hemorrhage,
  * Moderate to severe hepatic impairment,
  * Co-administration with a strong cytochrome P450 3A4 inhibitor (e.g. ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir),
* Other conditions at increased risk of bleeding:

  * Congenital or acquired coagulation disorder
  * Gastroduodenal bleeding within past 6 months,
  * Recent major trauma or surgery within past 30 days,
  * Concomitant use of fibrinolytics, oral anticoagulation, non-steroidal antiinflammatory drugs,
* Significant anemia,
* Increased risk of bradycardia,
* History of asthma or Chronic Obstructive Pulmonary Disease,
* Uric acid nephropathy,
* Ischemic stroke within 7 days,
* Heredity galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption,
* Concomitant use of a strong CYP3A4 inducer
* Concomitant use of CYP3A4 substrates with narrow therapeutic indices (e.g. cisapride, ergot alkaloids), simvastatin at a dose greater than 40 mg/d,
* Concomitant use of Selective Serotonin Reuptake inhibitors,
* Concomitant use of digoxin without close clinical and laboratory monitoring,
* Contra-indication to use Aspirin,
* Breast-feeding,
* Pregnancy,
* Adult protected by the law,
* Patient participating in another biomedical research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-11; Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
area under the curve corresponding to troponin level as a function of time | up to 24 hours
  Troponin kinetics during the first 24 hours following rotational atherectomy.

SECONDARY OUTCOMES:
area under the curve corresponding to troponin level as a function of time | up to 36 hours
Frequence of clinical events during the in-hospital period | One day before the procedure until 36 hours after.
  * Major life-threatening bleeding
  * Minor bleeding leading to clinically significant disability
  * Death from any cause,
  * Acute coronary syndrome with or without ST elevation,
  * Ischemic stroke,
  * In-stent thrombosis,
  * Coronary dissection or perforation,
  * Bail-out requiring anti GPIIb-IIIa administration.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Didier, PHD, Principal Investigator — University Hospital, Toulouse
Locations (4):
- France (4):
  - Clinique Pasteur, Toulouse, Haute-Garonne
  - Fédération de Cardiologie CHU TOULOUSE, Toulouse, Haute-Garonne
  - Hospices civils de Lyon, Lyon
  - University Hospital, Nîmes

REFERENCES:
- [Result] Lhermusier T, Motreff P, Bataille V, Cayla G, Farah B, Roncalli J, Elbaz M, Boudou N, Campello-Parada F, Bouisset F, Souteyrand G, Berard E, Bongard V, Carrie D. TIcagrelor in Rotational Atherectomy to Reduce TROPonin Enhancement: The TIRATROP Study, A Randomized Controlled Trial. J Clin Med. 2023 Feb 11;12(4):1445. doi: 10.3390/jcm12041445. PMID 36835980